CLINICAL TRIAL: NCT06571422
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of WJ47156 Monotherapy and in Combination With Other Anti-Tumor Therapies in Patients With Advanced Malignant Solid Tumors
Brief Title: Phase I Study of WJ47156 Monotherarpy and in Combination With Other Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS125-001-I
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-10

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- WJ47156 (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: WJ47156
- WJ47156+JS001+Bevacizumab (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: JS001+Bevacizumab
- WJ47146+JS207 (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: JS207

INTERVENTIONS:
Drug: WJ47156 — Monotherapy study: participate will recepit WJ47156 monotherpy with 3 dose groups; Combination therapy study: participate will recepit WJ47156 and other study drug if in the combination therapy period
  Arms: WJ47156
Drug: JS001+Bevacizumab — Participants in Cohort1 of combination therapy phase will receive WJ47156 plus toripalimab and bevacizumab.Toripalimab and bevacizumab are administered intravenously.
  Other Names: Toripaliman injection+Bevacizumab Injection
  Arms: WJ47156+JS001+Bevacizumab
Drug: JS207 — Participants in Cohort2 of combination therapy phase will receive WJ47156 plus JS207. JS207 is administered intravenously.
  Arms: WJ47146+JS207

SUMMARY:
This study is an open-label, dose-escalation and expansion, Phase I clinical study to evaluate the safety, tolerability, PK characteristics and preliminary antitumor activity of WJ47156 monotherapy and in combination with toripalimab in patients with advanced malignant solid tumors. The study consists of two parts, including monotherapy (Part 1) and combination therapy (Part 2).

ELIGIBILITY:
Inclusion criteria:

1. Male or female, 18 to 75 years old (inclusive) at the time of signing the ICF;
2. Patients with histologically or cytologically confirmed advanced malignant solid tumors；
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
4. Life expectancy ≥ 12 weeks;
5. At least one measurable lesion according to RECIST 1.1;
6. Adequate organ function ；
7. Female or male patients of childbearing potential must agree that they have no intention to become pregnant during the study and for 6 months after the last dose, and to use highly effective contraceptive methods with their partners; );
8. Voluntary participation with full informed consent by signing an written informed consent, and with good compliance.

Exclusion Criteria

1. CNS metastasis；
2. Pleural effusion, peritoneal effusion or pericardial effusion with clinical symptoms or requiring repeated treatment (e.g., puncture or drainage);
3. Unable to swallow tablets, intestinal obstruction, or other factors affecting the administration and gastrointestinal absorption of tablets
4. For the combination therapy, patients will not be enrolled in this study if they meet any of the following criteria:

（1）Imaging findings at screening showing tumor encasement of a major vessel or significant necrosis and cavity, which may lead to a hemorrhagic risk as judged by the investigator; （2）Patients with active autoimmune diseases requiring systemic treatment (e.g., corticosteroids or immunosuppressive drugs) within 2 years prior to the first dose, including but not limited to systemic systemic lupus erythematosus, multiple sclerosis, rheumatoid arthritis, inflammatory bowel disease, vasculitis, etc. However, hypothyroidism, hypoadrenalism or hypopituitarism controlled only by hormone replacement therapy, Type I diabetes mellitus not requiring systemic treatment, psoriasis or vitiligo are allowed; （3）Previously treated with anti-PD-1/L1 therapy; （4）History of interstitial lung disease or previous history of non-infectious pneumonia treated with corticosteroids, or evidence of active pneumonia on imaging at screening; （5）Gastrointestinal perforation, fistula, abdominal abscess and ulcerative disease or history of digestive system ulcerative disease within 6 months prior to the first dose (patients with stable ulcer as assessed by the investigator may be considered for enrollment); （6）Presence of serious, unhealed, or open wounds, active ulcers, or untreated fractures; （7）History of gastrointestinal bleeding within 6 months prior to enrollment, or clear tendency of gastrointestinal bleeding (including hemorrhagic risk of severe esophageal-gastric varices, locally active digestive tract ulcerative lesion, and persistent positive fecal occult blood); （8）Clinically significant hemoptysis or tumor bleeding for any reason within one month prior to the first dose; （9）History of obvious bleeding tendency or severe coagulation dysfunction; （10）Severe drug-related adverse events leading to permanent discontinuation of the drug product or bevacizumab or its analogues; （11）Use of antiplatelet therapy or anticoagulant therapy for treatment within 14 days prior to the first dose; （12）Long-term treatment with nonsteroidal anti-inflammatory drugs is permitted for brief periods of time to relieve symptoms such as fever or pain.

5. Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure > 100 mmHg) or history of hypertensive crisis or hypertensive encephalopathy; 6. Severe cardiovascular disease, including but not limited to, myocardial infarction, severe/unstable angina, congestive heart failure (New York Heart Association [NYHA] class ≥ 2), clinically significant supraventricular or ventricular arrhythmia requiring drug intervention, aortic aneurysm requiring surgical repair, any arterial thrombosis/embolism event, Grade 3 or higher (Common Terminology Criteria for Adverse Events [CTCAE] v5.0) venous thrombosis/embolism event, transient ischemic attack, cerebral vascular accident; Left ventricular ejection fraction (LVEF) < 50% by echocardiography. Corrected QT interval (QTc) > 480 ms (calculated using the Fridericia method; if QTc is abnormal, measure 3 times at an interval of 2 minutes and use the average).

7. Serious infection (CTCAE Grade > 2) within 28 days prior to the first dose, such as serious pneumonia, bacteremia, infection and complications requiring hospitalization; or active infection or unknown cause of fever (>38.5℃) requiring systemic anti-infection treatment within 2 weeks prior to the first dose (as judged by the investigator, patients with tumor-induced fever can be enrolled);

8. Presence of active tuberculosis, hepatitis B (positive for hepatitis B surface antigen [HBsAg] and HBV DNA higher than the lower limit of detection in the study site), hepatitis C (positive for HCV antibody [HCVAb] and HCV RNA higher than the lower limit of detection in the study site);

9. History of immunodeficiency, including human immunodeficiency virus (HIV) positive test, or history of known allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;

10. History of another primary malignant tumor, with the exception of malignant tumors (e.g., basal cell carcinoma of skin and squamous cell carcinoma of skin) who have received potentially curative therapy (more than 5 years) without known active disease prior to the first dose, without potential risk for recurrence ;

11. Toxicity of previous antitumor therapy has not been recovered to CTCTAE Grade ≤ 1 or to the level specified in the inclusion/exclusion criteria, with the exception of the following: related toxicities that are well controlled as judged by the investigator and do not affect the safety and compliance of the study treatment, and can be screened after confirmation by the Sponsor;

12. Prior use of the following drugs or therapies before the first dose:

1. Having received chemotherapy, immunotherapy or other anti-tumor therapy or other investigational drug within 21 days prior to the first dose, or having received oral fluorouracil, small-molecule targeted drugs or Chinese herbal products for antitumor indications within 14 days prior to the first dose;
2. Major surgery, radiation therapy (with the exception of palliative radiation to a localized bone or brain lesion, which may be completed up to 14 days prior), or any other minor surgical procedure, excluding placement of vascular access devices, within 28 days prior to the first dose; and any biopsy or other minor procedure within 7 days prior to the first dose.
3. In the combination therapy phase, patients who have received systemic treatment with corticosteroids (more than 10 mg/day prednisone or equivalent) or other immunosuppressants within 2 weeks prior to the first dose are allowed to use inhaled or topical steroids or systemic prednisone ≤10 mg/day and equivalent drug product;
4. Having received any live vaccine or attenuated live vaccine within 28 days prior to the first dose or requiring to be vaccinated with live vaccine or attenuated live vaccine during the study (only for patients in combination therapy phase);

   13. Patients who, in the opinion of the investigator, may be at increased risk of participation in the study due to other serious physical or mental diseases or abnormal laboratory examination, or may affect the compliance with treatment or interfere with the study results, and are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
1.DLT | 1 years
  Safety endpoints: incidence and severity of DLT
2、AE | 2.5 years
  Safety endpoints: incidence and severity of adverse events (AE); Abnormal changes in laboratory and other tests with clinical significance
3、SAE | 2.5 years
  Safety endpoints: incidence and severity of serious adverse events (SAE); Abnormal changes in laboratory and other tests with clinical significance
4.MTD | 1 year
  Maximum tolerated dose (MTD)
5.RP2D | 1 year
  Recommended dose for phase II trial

SECONDARY OUTCOMES:
6.ORR | 2 years
  Efficacy endpoints: Objective response rate (ORR) per RECIST v1.1
7.DOR | 2 years
  Efficacy endpoints: Duration of response (DOR) per RECIST v1.1
8.DCR | 2 years
  Efficacy endpoints: Disease control rate (DCR) per RECIST v1.1
9.PFS | 2 years
  Efficacy endpoints: Progression-free survival (PFS) per RECIST v1.1
10.OS | 2.5 years
  Efficacy endpoints: Overall survival (OS)
11.Peak concentration（Cmax） | 2 years
  The pharmacokinetic parameters of WJ47156：peak concentration (Cmax)
12.The time to receive Cmax（Tmax） | 2 years
  The pharmacokinetic parameters of WJ47156 ：the time to receive Cmax（Tmax）
13. Area under the plasma concentration-time curve (AUC0-t, AUC0-∞) | 2 years
  The pharmacokinetic parameters of WJ47156 ：area under the plasma concentration-time curve (AUC0-t, AUC0-∞)
14.Apparent volume of distribution (Vd/F) | 2 years
  The pharmacokinetic parameters of WJ47156 ：apparent volume of distribution (Vd/F)
15.Apparent clearance (CL/F) | 2 years
  The pharmacokinetic parameters of WJ47156 ：apparent clearance (CL/F)
16.Terminal half-life (t1/2) | 2 years
  The pharmacokinetic parameters of WJ47156 ：terminal half-life (t1/2)
17.Steady-state peak concentration(Cmax,ss) | 2 years
  The pharmacokinetic parameters of WJ47156 ：steady-state peak concentration(Cmax,ss) for the main PK parameters for multiple dose
18.Plasma trough concentration at steady state(Cmin,ss) | 2 years
  The pharmacokinetic parameters of WJ47156 ：Plasma trough concentration at steady state(Cmin,ss) for the main PK parameters for multiple dose
19.Mean plasma concentration at steady state(Cav,ss) | 2 years
  The pharmacokinetic parameters of WJ47156 ：mean plasma concentration at steady state for the main PK parameters for multiple dose
20.The time to receive Cmax at steady state（Tmax,ss） | 2 years
  The pharmacokinetic parameters of WJ47156 ：the time to receive Cmax at steady state（Tmax,ss）for the main PK parameters for multiple dose)
21.Area under the plasma concentration-time curve at steady state (AUC0-t, ss) | 2 years
  The pharmacokinetic parameters of WJ47156 ：area under the plasma concentration-time curve at steady state (AUC0-t, ss)for the main PK parameters for multiple dose)
22.Accumulation factor(RAC) | 2 years
  The pharmacokinetic parameters of WJ47156 ：accumulation factor(RAC) at steady state for the main PK parameters for multiple dose)
23.Fluctuation coefficient(FD) | 2 years
  The pharmacokinetic parameters of WJ47156 ：fluctuation coefficient(FD) at steady state for the main PK parameters for multiple dose)

OTHER OUTCOMES:
QT interval | 2 years
  To evaluate the correlation between plasma concentration of WJ47156 and QT interval (only applicable to the dose group of 30 mg and above of WJ47156 monotherapy)
Anti-drug antibody (ADA) | 2 years
  To evaluate the immunogenicity of toripalimab and JS207, including the incidence and titer of anti-drug antibody (ADA), if ADA positive, the neutralizing antibody (Nab) as needed
Blood concentration | 2 years
  Blood concentration of toripalimab and JS207

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No